CLINICAL TRIAL: NCT02688543
Title: Analgesic Effect and Functional Improvement Caused by Radiofrequency Ablation of Genicular Nerves in Patients With Advanced Osteoarthrosis of the Knee Joint Until 1 Year Following Treatment
Brief Title: Radiofrequency Ablation of Genicular Nerves for Advanced Osteoarthrosis of the Knee Joint 1 Year Follow-up.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General de Jerez de la Frontera (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RF knee 001
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Painful Osteoarthritis of the Knee
Keywords: radio frequency treatment; genicular nerves; osteoarthritis of the knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Radiofrequency Ablation; Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RF treatment (Experimental): Patients treated with radio frequency of the genicular nerves
  Interventions: Procedure: RF treatment; Radiation: radiofrequency ablation; Device: ultrasound

INTERVENTIONS:
Procedure: RF treatment — the genicular nerves are identified with the help of landmarks, ultrasound and nerve stimulation. Once the needle is correctly placed high frequency current is passed through the probe during 90 seconds at 20 V with tip temperature put to 80°C.
Radiation: radiofrequency ablation
Device: ultrasound

SUMMARY:
Pharmacological treatment of pain due to osteoarthritis of the knee often proves to be inadequate and/or cause intolerable side effects. Arthroplasty of the knee may offer a solution, but waiting lists may be long or certain patients may not be apt for a surgical intervention. Therefore an alternative pain treatment that is effective and has little side effects allowing to offer pain relief to those difficult to manage patients would be an added value in the therapeutic options.

We studies the short and long-term effects of radio frequency treatment of the genicular nerves in patients with severe pain due to osteoarthritis of the knee.

DETAILED DESCRIPTION:
Radio frequency treatment (RF) of the genicular nerves was found to be effective in a randomized controlled trial. Because of the blinding patients were allowed to continue pre-intervention pharmacological treatment, which may have interfered with the outcome. The short follow-up (12 weeks) does not allow drawing conclusion on the duration of the effect.

We aimed at assessing the pain reducing effect of RF of the genicular nerves and the duration of the effect.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from pain caused by osteoarthrosis of the knee joint
* osteoarthrosis of the knee joint (grade 3-4 according to the Kellgren Lawrence classification)
* pain of moderate to severe intensity (VAS≥5, on a 10-point scale) during >3 months
* pain resistant to conservative treatments

Exclusion Criteria:

* acute knee pain associated with radicular neuropathy or intermittent claudication, connective tissue diseases affecting the knee, serious neurologic or psychiatric disorders, mental deterioration impeding adequate communication or collaboration, injection with steroids or hyaluronic acids during the previous 3 months, anticoagulant medications, pacemakers, and prior electro-acupuncture treatment

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Pain reduction | 1, 6 and 12 months
  Pain intensity is measured using a 10-point VAS score

SECONDARY OUTCOMES:
Global patient satisfaction | 1,6 and 12 months
  Satisfaction is scored on a 4-point Likert scale: 1 (poor), 2 (average), 3 (good) and 4 (very good)
Improvement of quality of life | 1,6 and 12 months
  evaluated using the Western Ontario and MacMaster Universities Index of Osteoarthrosis (WOMAC)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General de Jerez de la Frontera (Servicio Andaluz de Salud), Jerez de la Frontera, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santana Pineda MM, Vanlinthout LE, Moreno Martin A, van Zundert J, Rodriguez Huertas F, Novalbos Ruiz JP. Analgesic Effect and Functional Improvement Caused by Radiofrequency Treatment of Genicular Nerves in Patients With Advanced Osteoarthritis of the Knee Until 1 Year Following Treatment. Reg Anesth Pain Med. 2017 Jan/Feb;42(1):62-68. doi: 10.1097/AAP.0000000000000510. PMID 27875368